CLINICAL TRIAL: NCT06454747
Title: A Randomized, Observer-Blinded, Placebo-Controlled Study on the Safety and Efficacy of Twice Daily Application of SM-030 Gel 0.64% Vs. SM-030 Gel 0.08% Vs. Placebo Gel in Adults With Melasma
Brief Title: Randomized Study Using SM-030 Gel for Adults With Melasma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-214
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: Randomized 3-arm tranche of main cohorts
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SM-030 gel 0.64% (Experimental): Topical application of SM-030 gel 0.64% twice daily for 12 weeks and a 4-week additional safety follow-up period.
  Interventions: Drug: SM-030 gel 0.64%
- Placebo gel (Placebo Comparator): Inactive comparator.
  Interventions: Drug: Placebo gel
- SM-030 gel 0.08% (Experimental): Topical application of SM-030 gel 0.08% twice daily for 12 weeks and a 4-week additional safety follow-up period.
  Interventions: Drug: SM-030 gel 0.08%

INTERVENTIONS:
Drug: SM-030 gel 0.64% — Topical application to face twice daily for 12 weeks.
  Arms: SM-030 gel 0.64%
Drug: Placebo gel — Topical application to face twice daily for 12 weeks.
  Arms: Placebo gel
Drug: SM-030 gel 0.08% — Topical application to face twice daily for 12 weeks.
  Arms: SM-030 gel 0.08%

SUMMARY:
Brief Summary This is a phase 2b, observer-blinded, randomized study that will evaluate the safety and efficacy of topically applied SM-030 gel 0.64% and SM-030 gel 0.08% compared against placebo gel in healthy adult male and female subjects with Melasma. The study will be comprised of a 12-week twice daily dosing period and a 4-week additional safety follow-up period. Approximately 138 subjects who meet the eligibility criteria, notably with a clinical diagnosis of Melasma will be randomized in a 3:2:1 ratio to one of three treatment arms: SM-030 gel 0.64% (N=69), Placebo gel (N=46), or SM-030 gel 0.08% (N=23). Subjects will be competitively enrolled in Mexico and El Salvador across 5 sites (4 sites in Mexico and 1 in El Salvador). Subjects will be assessed for safety and efficacy at each visit.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in the study:

1. Subjects must meet all of the following criteria to be included in the study:
2. Male or Female age 18-65 with Fitzpatrick skin type II through V and a clinical diagnosis of Melasma
3. Subjects with moderate to severe Melasma using the following guidelines:

1. Stable (unchanged per subject reporting) melasma for at least 3 months 2. Macular lesions, neither depressed nor atrophic 3. Melasma Severity Score of at least 2 (hyperpigmentation at least moderately darker than surrounding normal skin 3. Ability to understand, agree to, and sign the study informed consent form (ICF).

4. For female or childbearing subjects, they must be on an agreeable form of birth control (oral contraceptive therapies, estrogen replacement therapies, other non-oral hormonal therapies, IUDs, be abstinent, or have a vasectomized partner) and who have not added and/or changed the method of birth control in the last 6 months, and have no intention of adjusting or changing the method of birth control 5. Agree to discontinue all agents used to treat hyperpigmentation, aging or exfoliate the skin during the course of the study. Makeup and moisturizers are permitted.

6. Agree not to change their sun exposure at work, home, or leisure and apply study supplied sunscreen daily.

7. Technical ability and willingness to apply Investigational product. 8. Willing to allow digital photos of treatment and comparison areas to be taken and stored.

9. Willing to apply study-supplied mineral sunscreen, moisturizer, and cleanser to the face daily throughout the duration of the study

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded in the study:

1. Positive urine pregnancy test, pregnant, lactating, or female of childbearing potential who does not agree to use an active method of birth control for the duration of the study.
2. Conditions at baseline that would interfere with evaluation of UV-tanned skin, especially other pigmentary disorders including, but not limited to vitiligo affecting the treatment and comparison sites.
3. Severe photodamage as assessed by the 10-point photo damage assessment scale (Griffiths et al., 1992); (McKenzie et al., 2011).
4. Presence of known concomitant diseases associated with the development of hyperpigmentation (e.g., thyroid, liver, adrenal).
5. Current tanning booth exposure or any kind of phototherapy within 3 months of Screening.
6. Current or past use of monobenzyl ether to depigment skin.
7. Use of the following topical preparations within a 28-day washout period: topical corticosteroids, topical bleaching products (hyroquinone, niacinamide, kojic acid, ascorbic acid, chemical peels, topical tranexamic acid (TXA)), UV light therapy and sunbathing, topical retinoids.
8. Use of the following systemic agents within the specified washout periods:

1. Systemic corticosteroids (28 days) 2. Systemic cyclosporine, interferon (6 months) 3. Systemic acitretin, etretinate, isotretinoin (6 months) 4. Systemic methotrexate (6 months) 5. Systemic tranexamic acid (TXA) 6. Systemic photoallergic, phototoxic, and or photosensitizing drugs (6 months including psoralens, sulfonamide drugs, tetracycline antibiotics, thiazide diuretics, phenothiazines, coal tar and derivatives, and tricyclic antidepressants, chlorpromazine, benoxaprofen, piroxicam, nalidixic acid, procainamide, phenytoin, antimalarial medications, some cystostatic agents)

9. Laser (ablative or non-ablative), microneedling, PRP, or light-based treatment of the treatment areas within 3 months of Screening.

10. Any dermatological conditions within the designated application area that could interfere with clinical evaluations or any disease state or physical condition which might expose the subject to an unacceptable risk by study participation (neurodermatitis, eczema, psoriasis, atrophy, rosacea, seborrheic dermatits, etc.).

11. Any underlying disease(s) or other dermatological conditions that require the use of exclusionary topical or systemic therapy (see Exclusion criteria 6, 7, and 8).

12. Known high daily exposure to the sun (>4 hours of sun exposure through work or daily activities) and/or frequent sunbathing/UV tanning.

13. Unwilling to discontinue applying any prescription or over the counter (OTC) topical product creams and ointments, other than makeup and moisturizers, on treatment area(s) at Baseline through their last day of study.

14. Treatment of any type of cancer within 6 months of Screening, with the exception of superficial skin cancers such as basal cell or squamous cell carcinoma outside of treatment area.

15. Known allergy to any of the Investigational product(s) or any components in the Investigational product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure.

16. Unable to meet the study attendance requirements.

17. Any history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol.

18. Participation in any other trial of an investigational drug or device within 30 days prior to enrollment or participation in a research study concurrent with this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Investigator Assessment of Global Improvement (IAGI) for subjects receiving SM-030 compared to placebo | 12 weeks after first dose
  Superiority of each Active over Placebo based on proportion of subjects with a lower Investigator Assessment of Global Improvement at Week 12 compared to Baseline. Minimum value 0 is best, or completely clear. Maximum value is 6, or worse and darker pigmentation.
Change in Investigator Assessment of Global Improvement (IAGI) for subjects receiving different SM-030 concentrations | 12 weeks after first dose
  Superiority of SM-030 gel 0.64% over SM-030 gel 0.08% based on proportion of subjects with a lower Investigator Assessment of Global Improvement at Week 12 compared to Baseline. Minimum value 0 is best, or completely clear. Maximum value is 6, or worse and darker pigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Daivd Zepeda, MD, Principal Investigator — Zepeda Dermatologia
Locations (2):
- El Salvador (2):
  - Zepeda Dermatologia, Santa Tecla, La Libertad Department
  - Centro de Investigación y Desarrollo Brioso Ramirez, Santa Tecla, La Libertad, El Salvador